CLINICAL TRIAL: NCT07186036
Title: The Effect of a Soft Lumbosacral Body Brace Supporting Physiological Lordosis on Postural Control and Walking Speed in Children With Cerebral Palsy
Acronym: Cerebral palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Asiya Uzun, Assistant Proffesor, Kahramanmaras Sutcu Imam University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ethics committee app: 2025/047
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy GMFCS-ER I-II
Keywords: cerebral palsy,; walking; postur; postural control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: In our study, a lordosis angle will be created to support the existing lordosis using a steel-baleen elastic soft lumbosacral orthosis, and its effect on performance will be investigated using the tests applied. A soft lumbosacral orthosis suitable for the individuals will be used in three dimensions. Half of the individuals will be evaluated using these test methods first with a corset and then without a corset; the other half will be evaluated first without a corset and then with a corset. Tests will be repeated before and after orthosis use to determine the effectiveness of the orthosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In our study, a lordosis angle will be created to support the existing lordosis using a steel-balee (Experimental): In our study, a lordosis angle will be created to support the existing lordosis using a steel-baleen elastic soft lumbosacral orthosis, and its effect on performance will be investigated using the tests applied. A soft lumbosacral orthosis suitable for the individuals will be used in three dimensions. Half of the individuals will be evaluated using these test methods first with a corset and then without a corset; the other half will be evaluated first without a corset and then with a corset. Tests will be repeated before and after orthosis use to determine the effectiveness of the orthosis.
  Interventions: Device: soft lumbosacral orthosis

INTERVENTIONS:
Device: soft lumbosacral orthosis — The effect of trunk corsets on postural control and walking, GYA independence

SUMMARY:
The aim of this study is to investigate the effect of soft lumbosacral body braces on postural control and walking speed in children with cerebral palsy.

Hypothesis 1: Soft lumbosacral orthoses that support physiological lordosis in children with cerebral palsy improve postural control. Hypothesis 1: Soft lumbosacral orthoses that support physiological lordosis in children with cerebral palsy correct posture. Hypothesis 2: A soft lumbosacral body corset increases walking speed in children with cerebral palsy.

The number of individuals to be included in the study has been determined using G*Power 3.1.9.7 effect size: 0.80, α = 0.05, power: 0.95. Individuals with CP who attend specific rehabilitation centres in Gaziantep and Kahramanmaraş and have GMFCS levels 1 and 2 will be included in the study. The necessary permissions will be obtained from the centres. The demographic information, clinical levels, and clinical types of the individuals will be recorded using a form. The Postural Control Measurement in Sitting, Paediatric Berg Balance Test, and Functional Reach Test will be used to assess the postural control of children with SP. Walking speed will be assessed using the Timed Up and Go Test. In our study, a lordosis angle will be created to support the existing lordosis using a steel-baleen elastic soft lumbosacral orthosis, and its effect on performance will be investigated using the tests applied. A soft lumbosacral orthosis suitable for the individuals will be used in three dimensions. Half of the individuals will be evaluated using these test methods first with a corset and then without a corset; the other half will be evaluated first without a corset and then with a corset. Tests will be repeated before and after orthosis use to determine the effectiveness of the orthosis.

ELIGIBILITY:
Inclusion Criteria:Children with cerebral palsy

* Aged 6-15 years
* GMFCS 1-2
* Voluntarily participating in the study

Exclusion Criteria:Children with cerebral palsy

* Inappropriate GMFCS level
* Presence of orthopaedic problems that may affect balance
* Lack of cooperation from the individual

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional Reach Test | The first day of assesment
  Developed by Duncan et al. in 1990 to assess dynamic balance. The maximum distance reached forward with the arm without disrupting the fixed standing position is measured. The distance between the third metacarpals is measured at the start and end positions of the test. The subject is asked to reach forward three times, and the average is taken. It is valid and reliable for children with SP (ICC = 0.94, 0.97, 0.98).
Seated Postural Control Measurement (SPCM) | The first day of assesment
  Developed by a team of occupational therapists and physiotherapists at Sunny Hill Health Centre in Vancouver, Canada, to assess seated posture. SPCM evaluates the child's postural impairment as well as the effect of sitting on postural control.
Paediatric Berg Balance Test | the first day of assesment
  The Paediatric Berg Balance Scale (PBBS), a version of the Berg Balance Scale adapted for children by Franjoine and colleagues, will be used to assess functional balance in daily living activities. The scale consists of 14 items, each scored from 0 to 4, with a maximum possible score of 56.
Timed Up and Go Test (TUG) | the first day of assesment
  Used to assess functional mobility and dynamic balance. The TUG is a valid and reliable test for assessing balance in children with cerebral palsy (r=0.99). A chair with a backrest but no armrests is used for the assessment. The test begins with the child sitting on the chair with their hips and knees flexed at 90°. The child is asked to stand up from the chair, walk 3 metres, and sit back down. The time taken from standing up from the chair to sitting back down is recorded. The test is repeated 3 times, and the average of these three values is taken for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam Üniversitesi, Kahramanmaraş, onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No